CLINICAL TRIAL: NCT07204379
Title: Effects of Three Oral Analgesics on Postoperative Pain Following Root Canal Preparation: a Controlled Clinical Trial
Brief Title: Effect of Oral Analgesics on Post-op Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Safina Habib, Principal investigator, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AFID Safeena
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — L 5409709; Tramadol; Naproxen

STUDY DESIGN:
Intervention Model Description: patients to be divided into 4 equal groups and different drugs to be administered amongst each group and efficacy evaluated afterwards.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo group (Placebo Comparator): this group to be administered placebo medication (multi-vitamins)
  Interventions: Other: No intervention?placebo
- Novafen group (Active Comparator): this group to be administered Novafen medication
  Interventions: Drug: Novafen
- Tramadol group (Active Comparator): this group to be administered Tramadol Medication
  Interventions: Drug: Tramadol
- Naproxen group (Active Comparator): this group to be administered Naproxen medication
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Novafen — Novafen analgesic medication to be administered as pain painkiller in one group of patients undergoing root canal therapy
  Arms: Novafen group
Drug: Tramadol — Tramadol analgesic medication to be administered as pain painkiller in one group of patients undergoing root canal therapy
  Arms: Tramadol group
Drug: Naproxen — naproxen analgesic medication to be administered as pain painkiller in one group of patients undergoing root canal therapy
  Arms: Naproxen group
Other: No intervention?placebo — multivitamins to be administered in this group
  Arms: Placebo group

SUMMARY:
after 2 visit endodontics treatment, the analgesic efficacy of three different medications will be evaluated.

DETAILED DESCRIPTION:
Patients will be divided randomly into four groups of 25 patients each a control group receiving a single dose of a placebo (multivitamines) and three experimental groups receiving either a single dose of a Tramadol tablet (100 mg of Tramadol hydrochloride) Novafen capsules [325 mg of paracetamol (acetaminophen)], 200 mg of ibuprofen and 40 mg of caffeine anhydrous) or Naproxen tablets (500 mg of naproxen) immediately on completion of the first appointment. Balanced block random allocation will be made (12 blocks contained eight patients and one block contained four patients) by generating random digits via Microsoft Excel 2007. An Assistant who will be blinded to the aim and the protocol of the study generated the numbers. After explanation of the treatment procedures, treatment will be performed under rubber dam isolation by the dentist. The tooth will be anaesthetized using one cartridge of Ligocaine HCL 2%with Adenaline 0.001% injection 1.8ml (Septodont) local anaesthetic solution. If pain still remained during access cavity preparation, intrapulpal anaesthesia will be used as supplementary anaesthesia. The investigator who performed the root canal treatment will be blinded to the assignment. An access cavity will be prepared, and the working length will be determined electronically using an apex locator (Dentaport ZX; J. Morita, MFG,CORP) 1 mm short of the apex with a size 15 or 20 K-file and confirmed by periapical radiographs. The apical part of each root canal will be prepared to a size 25 K-file with the step- back technique in a circumferential manner. Normal saline (sodium chloride B.P0.9%W/V IV Infusion (sterifluid NS))will be used as the irrigant solution between each instrument. Canals will then be dried with paper points, and the access cavities will be restored temporarily with Cavit (3M ESPE, St Paul, MN, USA). Each patient's tablet/ capsule will be inserted into a sealed coded packet by a trained person who will be blinded to the drugs, and the packet remained sealed until it will be given to the patient. The patients will be supervised by one of the investigators when taking the oral medications. The intensity of the preoperative pain will then be measured by instructing the patient to complete a Visual Analogue Scale (VAS) before treatment and after 6, 12 and 24 h. At the second appointment, 24 h later the root canal treatment will be completed. The markings on the VAS will be measured, and the degree of pain will be categorized as mild (scores 1-3), moderate (scores 4-6) or severe (scores 7-10).

ELIGIBILITY:
Inclusion Criteria:

1- Patients were aged between 20 and 60 years 2. Patients with moderate to severe spontaneous pain associated with irreversible pulpitis in single-rooted 3- premolars or anterior teeth with no clinical or radiographic signs or symptoms of acute or chronic apical periodontitis

Exclusion Criteria:

1. Systemic disease
2. Pregnant womens
3. History of taking analgesics in previous 12 hrs or other drugs prior to presenting for treatment.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Post operative pain | 6 hours - 72 hours
  Post operative pain to be measured/evaluated in patients undergoing root canal therapy using visual analog scale (VAS). This is a numeric scale with readings 0-10. with 0 indicating no pain, 1-3 indicating mild pain, 4-6 indicating moderate pain, and 7-10 indicating severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- AFID, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No